CLINICAL TRIAL: NCT02878109
Title: Dynamic Contrast-enhanced Magnetic Resonance Imaging for Assessment of Response to Transarterial Chemoembolization of Hepatocellular Carcinoma
Brief Title: DCE-MRI for Assessment of Response to TACE of HCC
Acronym: DCE-MRI
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Other Study IDs: CE15.388
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2018-01

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Magnetic resonance imaging (MRI); Transarterial chemoembolization (TACE)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Post-treatment phase group: 29 patients will undergo: 4D-THRIVE and 4D-FLOW sequences during magnetic resonance imaging (MRI) before and after transarterial chemoembolisation (TACE).
  Interventions: Device: Post-treatment phase group
- Pre-treatment phase group: 11 patients will undergo: 4D-THRIVE and 4D-FLOW sequences during magnetic resonance imaging (MRI) before treatment (if any).
  Interventions: Device: Pre-treatment phase group

INTERVENTIONS:
Device: Post-treatment phase group — 4D-THRIVE and 4D-FLOW using magnetic resonance imaging (MRI)
  Groups: Post-treatment phase group
Device: Pre-treatment phase group — 4D-THRIVE and 4D-FLOW using magnetic resonance imaging (MRI)
  Groups: Pre-treatment phase group

SUMMARY:
This study is conducted to evaluate dynamic contrast-enhanced MRI to quantify the efficacy of trans-arterial chemoembolization by comparing imaging results before and after treatment for at least one hepatic tumor and to look at blow flow curves of the free-breathing MRI before treatment.

DETAILED DESCRIPTION:
Background: Liver cancer is the second leading cause of cancer deaths worldwide. Hepatocellular carcinoma (HCC) typically presents arterial phase hyperenhancement. For intermediate stage disease and the majority of patients not eligible for curative therapies, transarterial chemoembolization (TACE) is considered as the first-line palliative treatment in eligible patients.

Despite its efficacy on HCC, TACE presents major challenges such as the lack of quantitative biomarkers of treatment response. Dynamic contrast-enhanced MRI (DCE-MRI) enables quantitative assessment of tumor and tissue enhancement, by acquiring MR signal intensity as a function of time.

Objectives: This study is conducted: 1) to develop a monitoring system based on quantifiable measures during intra-arterial treatments from dynamic MRI, using time-activity curves analyzed using a dual-input dual-compartment model, and 2) to look at blood flow curves of the MRI before the treatment, if any, for at least one tumor, without requiring any breath hold.

Design:

* Post-treatment phase group: This will be a prospective study in HCC patients undergoing TACE (including DC beads) according to their clinical standard of care. A 4D-THRIVE sequence will be performed. Single intensities before/after gadolinium-based contrast agent enhancement will be used to create time-concentration curves, which will be fitted to a simple perfusion model that accounts for the dual blood supply of the liver through the hepatic artery and the portal vein. Perfusion parameters of arterial hepatic blood flow, portal venous hepatic blood flow, total hepatic blood flow and arterial fraction will be extracted from the model and compared between HCC and surrounding cirrhotic liver. When deemed necessary, a CBCT can be acquired before chemo-embolization in way to see that the appropriate artery is selected for the treatment. The CBCT will be used when available to determine the parameters of the blood flow obtained with our model.
* Pre-treatment phase group: This will be a prospective study in HCC patients undergoing a MRI according to their clinical standard of care. A 4D-THRIVE sequence will be performed. Single intensities before/after gadolinium-based contrast agent enhancement will be used to create time-concentration curves, which will be fitted to a simple perfusion model that accounts for the dual blood supply of the liver through the hepatic artery and the portal vein. Perfusion parameters of arterial hepatic blood flow, portal venous hepatic blood flow, total hepatic blood flow and arterial fraction will be extracted from the model and compared between HCC and surrounding cirrhotic liver.
* Comparison: A comparison between the blood flow curves between the post-treatment phase group [apnea] and the pre-treatment phase group [free-breathing] will be done.

Methods: Forty patients will be selected. For twenty-nine of them [post-treatment phase group], a 4D-THRIVE sequence will be acquired within 2 weeks prior to TACE and between 6 and 8 weeks after TACE. A 4D-FLOW MRI sequence will also be included. For the remaining eleven patients [pre-treatment phase group], only a 4D-THRIVE sequence will be acquired within 2 weeks prior to treatment, if any, including a 4D-FLOW MRI sequence.

Expected results: The results of this study will provide quantitative DCE-MRI biomarkers for identification of viable tumor and tumor response. In addition, presence of increased % arterial flow and decreased portal venous flow in HCC using DCE-MRI are expected to help to assess treatment response.

ELIGIBILITY:
Inclusion Criteria:

* All patients:

  * Are at least 18 years old at screening;
  * Able to comprehend and willingness to provide voluntary consent;
  * Have at least one HCC;
  * HCC lesion of at least 10 mm;
  * Understand French or English instruction.
* Post-treament phase group:

  * Are able to have a MRI before and after TACE;
  * Must undergo a TACE as part of their clinical standard of care for HCC;
  * Have a new prescription for TACE for at least one HCC.
* Pre-treatment phase group:

  * Are able to have a MRI before treatment (if any);
  * Must undergo an MRI as part of their clinical standard of care for HCC.

Exclusion Criteria:

* Have any contra-indication for MRI (such as claustrophobia, pacemaker, metallic clips for a neurosurgical procedure);
* Are pregnant or trying to become pregnant;
* Have a weight or girth preventing them from entering the MR magnet bore;
* Are unable to understand or unwilling to provide written informed consent for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is adults with a hepatocellular carcinoma (HCC). The post-treatment phase group will also encompass patients with a planned transarterial chemoembolization (TACE). For the purpose of this study, the investigators will recruit patients who will be treated at the CHUM.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Hepatic and tumor blood flow before and after TACE | Within 2 weeks before TACE and 6 to 8 weeks after TACE
  Measures of hepatic and tumor blood flow will help in describing HCC angiogenesis and in determining the efficiency of TACE on the tumor.
Hepatic and tumor blood flow before HCC treatment | Within 2 weeks before HCC treatment
  Measures of hepatic and tumor blood flow will help in describing HCC angiogenesis

CONTACTS AND LOCATIONS:
Overall Officials: An Tang, MD, MSc, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal, Montreal, Quebec, Canada